CLINICAL TRIAL: NCT01240499
Title: Intervention s'Inspirant du Nouveau Paradigme en matière de Gestion de Poids Chez Des Femmes préménopausées présentant un Surplus de Poids
Brief Title: Effects of a Health-At-Every-Size Approach on Weight Management in Premenopausal Overweight Women
Acronym: CHOIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Simone Lemieux, Professeur, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHOIX-170
Record Dates: First submitted 2010-11-09; First posted 2010-11-15 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Overweight
Keywords: Weight management; New weight paradigm; Overweight women; Eating behaviors; Appetite ratings; Blood lipids
MeSH Terms: conditions — Overweight; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Health-At-Every-Size (HAES) (Experimental)
  Interventions: Other: Health-At-Every-Size (HAES)
- Social Support (SS) (Active Comparator)
  Interventions: Other: Health-At-Every-Size (HAES)
- Control (No Intervention)

INTERVENTIONS:
Other: Health-At-Every-Size (HAES) — 1. HAES group: 14 weekly sessions.
     Focus on general well-being and positive ways of having a healthy and satisfying lifestyle. Supported by lectures, guided self-reflection, group discussions, as well as practical exercises, this intervention aims at enhancing awareness and knowledge about biological, psychological, and sociocultural aspects of body weight.
  2. SS group: 14 weekly sessions.
  The objective is to reproduce a structural social support provided by the group itself. Each participant offers their support to each other. Each theme discussed in the HAES group is repeated in the SS group but the health professionals in charge of the group (dietitian & psychologist) are not counselors (as in HAES group) but only facilitators.
  Outcome measures: For all women under study.
  Other Names: Non applicable
  Arms: Health-At-Every-Size (HAES); Social Support (SS)

SUMMARY:
The purpose of this study is to measure the effects of a Health-At-Every-Size (HAES) approach on global health status of premenopausal overweight women preoccupied about their weight and who have been unsuccessful in previous weight loss attempts.

DETAILED DESCRIPTION:
Weight management is a critical issue in developed countries where the prevalence of obesity is increasing. Poor long-term success observed with current weight-control strategies stresses the relevance to explore new weight management approaches. One of these approaches, referred to as Health-At-Every-Size (HAES), is a new weight paradigm that focuses on a healthy lifestyle by promoting overall health benefits of behavioral changes related to dietary habits and physical activity and emphasizes self-acceptance and well-being, independently of body weight status. Studies on the effects of a HAES approach have shown significant improvements in metabolic and psychological variables.

To our knowledge, no study has yet reported the short and long-term impacts of a HAES approach on a cluster of variables (psychological, morphological, metabolic, and nutritional) in women. The aim of this study is to measure the effects of a HAES approach on global health status of premenopausal overweight women preoccupied about their weight and who have been unsuccessful in previous weight loss attempts. In this parallel controlled trial, women will be randomized to one of the 3 treatment conditions: HAES group, Social support group (SS), or Control group. Measurements will be taken in the short term as well as in the long term (up to 1 year post-intervention).

ELIGIBILITY:
Inclusion criteria:

* Healthy premenopausal women from Quebec City metropolitan area
* Age: between 30 to 50 years old
* Stable body weight (+/- 2 kg) for at least 2 months before the beginning of the study
* Overweight or obesity: Body mass index [BMI] between 25 and 35 kg/m2
* Preoccupation about weight and eating: showing overconcern with shape and weight, exhibiting restriction over food choices for at least 2 years, and having been unsuccessful in previous attempts to lose weight (for at least the past 2 years)
* Current weight corresponding to maximum weight reached during adult lifetime

Exclusion criteria:

* Women currently dieting to lose weight
* Taking oral contraceptives or postmenopausal status
* Pregnant or lactating women
* Under treatment for coronary heart disease, diabetes, dyslipidemia, hypertension, depression or endocrine disorders (with the exception of stable thyroid disease)
* Women presenting metabolic or important psychological disorders (drug or alcohol abuse, bulimia, …)
* Women who had already take part to the Health-At-Every-Size (HAES) approach

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2003-09; Primary Completion 2006-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in global health status outcomes (metabolic, psychological and nutritional variables, physical activity habits) from baseline to the end of the intervention, and at 6 and 12 months post-intervention. | At baseline and at the end of the intervention period (4 months), and at 6 months and 1 year post-intervention (10 months and 16 months, respectively).
  Plasma LDL-cholesterol concentrations, Eating behaviors (restraint, disinhibition, and susceptibility to hunger), appetite ratings (desire to eat, hunger, fullness, and prospective food consumption), psychological variables (e.g. quality of life, self-esteem), physical activity habits, dietary intakes.

SECONDARY OUTCOMES:
Anthropometric and metabolic variables | At baseline and at the end of the intervention period (4 months), and at 6 months and 1 year post-intervention (10 months and 16 months, respectively).
  Anthropometric measures (body mass index, waist and hip circumferences) and metabolic variables (blood lipids, insulin and glucose levels, blood pressure, resting metabolic rate, salivary cortisol levels).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lemieux, Ph.D., Dt.P., Principal Investigator — Department of food sciences and nutrition/Institute of Nutraceuticals and Functional Foods (INAF), Laval University
Locations (1):
- INAF, Laval University, Québec, Quebec, Canada

REFERENCES:
- [Result] Gagnon-Girouard MP, Begin C, Provencher V, Tremblay A, Boivin S, Lemieux S. Subtyping weight-preoccupied overweight/obese women along restraint and negative affect. Appetite. 2010 Dec;55(3):742-5. doi: 10.1016/j.appet.2010.09.011. Epub 2010 Sep 17. PMID 20851157
- [Result] Gagnon-Girouard MP, Begin C, Provencher V, Tremblay A, Mongeau L, Boivin S, Lemieux S. Psychological Impact of a "Health-at-Every-Size" Intervention on Weight-Preoccupied Overweight/Obese Women. J Obes. 2010;2010:928097. doi: 10.1155/2010/928097. Epub 2010 Jun 29. PMID 20798861
- [Result] Provencher V, Begin C, Tremblay A, Mongeau L, Corneau L, Dodin S, Boivin S, Lemieux S. Health-At-Every-Size and eating behaviors: 1-year follow-up results of a size acceptance intervention. J Am Diet Assoc. 2009 Nov;109(11):1854-61. doi: 10.1016/j.jada.2009.08.017. PMID 19857626
- [Result] Gagnon-Girouard MP, Begin C, Provencher V, Tremblay A, Boivin S, Lemieux S. Can we apply the dual-pathway model of overeating to a population of weight-preoccupied overweight women? Int J Eat Disord. 2009 Apr;42(3):244-52. doi: 10.1002/eat.20614. PMID 19034910
- [Result] Provencher V, Begin C, Gagnon-Girouard MP, Tremblay A, Boivin S, Lemieux S. Personality traits in overweight and obese women: associations with BMI and eating behaviors. Eat Behav. 2008 Aug;9(3):294-302. doi: 10.1016/j.eatbeh.2007.10.004. Epub 2007 Nov 6. PMID 18549988
- [Result] Provencher V, Begin C, Gagnon-Girouard MP, Gagnon HC, Tremblay A, Boivin S, Lemieux S. Defined weight expectations in overweight women: anthropometrical, psychological and eating behavioral correlates. Int J Obes (Lond). 2007 Nov;31(11):1731-8. doi: 10.1038/sj.ijo.0803656. Epub 2007 Jun 5. PMID 17549091
- [Result] Provencher V, Begin C, Tremblay A, Mongeau L, Boivin S, Lemieux S. Short-term effects of a "health-at-every-size" approach on eating behaviors and appetite ratings. Obesity (Silver Spring). 2007 Apr;15(4):957-66. doi: 10.1038/oby.2007.638. PMID 17426331
- [Derived] Leblanc V, Provencher V, Begin C, Corneau L, Tremblay A, Lemieux S. Impact of a Health-At-Every-Size intervention on changes in dietary intakes and eating patterns in premenopausal overweight women: results of a randomized trial. Clin Nutr. 2012 Aug;31(4):481-8. doi: 10.1016/j.clnu.2011.12.013. Epub 2012 Jan 31. PMID 22296874